CLINICAL TRIAL: NCT01887977
Title: Computational Modeling for Prediction of Acoustic Changes in Vowel Production
Brief Title: Computational Modeling for Prediction of Acoustic Changes in Vowel Production Due to Orthognathic Surgery
Acronym: PUMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: T17/2012
Record Dates: First submitted 2013-03-28; First posted 2013-06-27 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Jaw Deformity; Facial Asymmetry
Keywords: Orthognathic surgery; Speech production; MRI
MeSH Terms: conditions — Jaw Abnormalities; Facial Asymmetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Computational modeling (Experimental)
  Interventions: Other: MRI examination

INTERVENTIONS:
Other: MRI examination — The vocal and nasal tracts from the lips and nostrils to the beginning of the trachea are imaged with Siemens Avanto 1.5T MRI machine using carefully optimized, externally triggered imaging sequences that are synchronized with the rest of the experimental setting. A sound sample, given by the test subject, is recorded simultaneously to obtain a coupled data set: the speech sound and the precise anatomy which produces it.
  Other Names: with Siemens Avanto 1.5T MRI machine

SUMMARY:
A computational model of human sound production based on high quality anatomic measurements and physical laws of sound propagation cannot be accomplished without a comprehensive data set including both 3D-images of the speaker's anatomy and the simultaneous recording of speech. Since the computational model has separate models for the vocal folds and the vocal tract, patients undergoing an orthognathic surgery is an optimal test object for the model development. Vocal folds remain unchanged while substantial changes take place in the vocal tract. Moreover, since the aim of the research is to predict acoustic changes in speech due to operations in head neck area, the orthognathic patient group is par excellence an example of such a prediction problem. If the model can be shown to give valuable information pre-operationally, many other patient groups could benefit from the results.

DETAILED DESCRIPTION:
Orthognathic surgery deals with the correction of abnormalities of the facial tissues. The underlying cause for abnormality may be present at birth or acquired during the life as the result of distorted growth or trauma. Orthodontic treatment alone is not adequate in many cases due to severity of the deformities. In a typical operation, the position of either one jaw (mandible or maxilla) or both jaws is surgically changed in relation to the skull base. The movement of the jaw position varies usually between 5-15 mm either to anterior or posterior direction. Such a considerable movement has a very profound effect on the shape and volume of vocal tract resulting detectable changes in acoustics. Although the surgery involves mandibular and maxillary bone, changes occur also in the position and shape of respective soft tissues and hyoid bone, as well. For this project, 20 adult patients (10 women and 10 men) undergoing orthognathic surgery will be enrolled. Exclusion criteria include diseases and conditions in which MRI examination is contraindicated (.e.g. pace maker), severe speech or hearing impairment, and other situations where the patient has difficulties with completing the tasks defined in the research protocol. Furthermore, patients to whom segmental surgery of the jaws will be performed in connection of orthognathic surgery are excluded. A specific pre-selection criterion for patients is the presence of numerous dental amalgam fillings that may cause artifacts in MR images.

ELIGIBILITY:
Inclusion Criteria:

- Healthy patients undergoing orthognathic surgery

Exclusion Criteria:

* Patients with conditions in which MRI examination is contraindicated (e.g. pace maker)
* Patients who require several operations or segmented jaw surgery
* Patients with cognitive impairment
* Patients with numerous dental amalgam fillings that may cause artifacts in MR images

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Acoustic changes in vowel production of hte patients duoe to orthognathic surgery | 6 and 30 weeks postoperatively
  a measurement of sound formants

SECONDARY OUTCOMES:
Anatomical changes in vocal tract due to orthognathic surgery | 6 and 30 weeks postoperatively
  changes in vocal track dimensions

CONTACTS AND LOCATIONS:
Overall Officials: Risto P Happonen, Professor, Principal Investigator — Turku University Hospital, Po. Box 52, FI-20521 Turku, Finland
Locations (1):
- Turku University Hospital, Turku, Finland